CLINICAL TRIAL: NCT03044535
Title: Mechanical Circulatory Support: Measures of Adjustment and Quality of Life
Brief Title: Mechanical Support Measures of Adjustment and QOL
Acronym: MCS A-QOL
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kathleen Grady, Professor of Surgery and Medicine, Feinberg School of Medicine at Northwestern University, Northwestern University
Other Study IDs: STU00201984; 1R01HL130502-01 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Quality of Life; Heart Failure; Cardiovascular Diseases
Keywords: quality of life; mechanical circulatory support
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Longitudinal assessment: Assessments will be performed pre-MCS, 3 months post-MCS and 6 months post-MCS. Participants in this group must be scheduled for MCS implant.
- Group 2: Cross-sectional assessment: A one-time assessment will be performed on participants who are post-MCS implant (between 3 months and 10 years post-implant). Participants in this group must already have an MCS device in place.

SUMMARY:
The purpose of this study is to develop a measurement system to assess adjustment to mechanical circulatory support (MCS) (also referred to as a ventricular assist device [VAD]) and health-related quality of life (HRQOL) in patients with advanced heart failure who receive a VAD. This investigators refer to this measurement system as Mechanical Circulatory Support: Adjustment and Quality of Life (MCS A-QOL).

DETAILED DESCRIPTION:
It is estimated that 5.1 million U.S. adults have heart failure, with an incidence of 825,000 new cases annually. The prevalence of heart failure is expected to increase by 46% from 2012 to 2030. Mechanical circulatory support (MCS) has been developed as a bridge to heart transplantation and as permanent support (i.e., destination therapy). MCS devices help the heart pump blood to the body. Left ventricular assist devices (LVADs), a type of MCS, support the left heart.

Health-related quality of life (HRQOL) is a very important outcome that advanced heart failure patients care about when making health care decisions, including when considering surgical treatment options, such as heart transplantation and mechanical circulatory support.

Currently available HRQOL questionnaires do not assess the unique burdens of MCS, such as changing power sources and driveline exit site dressings; safety precautions (e.g., no immersion in water, need for an MCS-trained caregiver); troubleshooting VAD alarms; and MCS-specific complications, often associated with frequent hospitalizations. Since these questionnaires do not focus on issues of concern to MCS patients, they lack sensitivity and precision to measure the potentially wide-ranging impact of MCS on HRQOL.

Guided by the investigators empirically supported MCS A-QOL conceptual model, the investigators will use state-of-the-science psychometric measurement methods to create "item banks" (sets of items that comprise carefully calibrated questions which define and quantify a common theme) from the investigators existing MCS A-QOL item pools (library of relevant items). Using calibrated item banks, the investigators will develop computer adaptive tests (CATs) and fixed-length short forms to reduce respondent burden and enhance measurement precision. The investigators will assess reliability, validity, responsiveness to change, and clinically important differences of MCS A-QOL measures.

ELIGIBILITY:
Group 1 Inclusion Criteria

1. Advanced heart failure patients accepted for, or scheduled for, primary (first time) implant of a continuous flow MCS device left (L)VAD
2. The continuous flow MCS device implant strategy can be a bridge to transplant, destination therapy, or bridge to recovery
3. Age >= 19 years and able to speak and understand English
4. Sufficient cognitive ability to provide self-report data on a computer touchscreen/standard computer and/or on paper-based forms with minimal assistance.
5. Willing to participate and able to give written informed consent

Group 1 Exclusion Criteria:

1. Scheduled for implant of a bi-VAD, right (R)VAD, or total artificial heart

Group 2 Inclusion Criteria:

1. Patient with a continuous flow MCS device left (L)VAD who is more than 3 months post-implant at the following intervals: 3, 6, 12, 18, 24, 30, 36, 42, 48 months and every 6 months thereafter. Note: patients can have had prior MCS devices.
2. The continuous flow MCS device, implant strategy can be a bridge to transplant, destination therapy, or bridge to recovery
3. Age >= 19 years and able to speak and understand English
4. Sufficient cognitive ability to provide self-report data on a computer touchscreen/standard computer and/or on paper-based forms with minimal assistance
5. Willing to participate and able to give written informed consent

Group 2 Exclusion Criteria:

1. Has a bi-VAD, right (R)VAD, or total artificial heart

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is enrolling patients with advanced heart failure who require Mechanical Circulatory Support (MCS) to help the heart pump blood.
Sampling Method: Non-Probability Sample
Enrollment: 895 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Creation of new MCS A-QOL item banks and short forms and validation of existing instruments | Longitudinally: baseline through 6 months post-MCS implant and cross-sectionally through 10 years post-MCS implant
  Psychometric measurement methods will be used to create new "item banks" (sets of items that comprise carefully calibrated questions which define and quantify a common theme) and short forms from our existing MCS A-QOL item pools (library of relevant items). Psychometric properties (e.g., reliability, validity, etc) of these new measures and existing instruments, some of them modified, will be evaluated, in order to provide evidence of their clinical utility for measuring adjustment to MCS and HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen L Grady, RN, PhD, Principal Investigator — Northwestern University; Elizabeth A Hahn, MA, Principal Investigator — Northwestern University
Locations (12):
- United States (12):
  - University of California, San Diego, La Jolla, California
  - University of California, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - St. Vincent Hospital, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Integris Health, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All published resources generated during the course of this work will be made available to other investigators upon request. Per study procedure, the investigators will respond to requests from other researchers to use de-identified data and make MCS A-QOL measurement system available to both researchers and clinicians for use.
  Data that were derived from the Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs) will only be shared per data sharing protocols.

REFERENCES:
- [Derived] Hahn EA, Allen LA, Cella D, Beiser DG, Denfeld QE, Kirklin J, Lindenfeld J, McIlvennan CK, Ruo B, Teuteberg J, Kiernan M, Klein L, Lee CS, Murks C, Rich J, Stehlik J, Walsh MN, Bedjeti K, Grady KL. Responsiveness validity for measures of adjustment to life with a left ventricular assist device: Findings from the MCS A-QOL study. JHLT Open. 2025 Apr 22;9:100269. doi: 10.1016/j.jhlto.2025.100269. eCollection 2025 Aug. PMID 40485994
- [Derived] Grady KL, Kallen MA, Beiser DG, Lindenfeld J, Teuteberg J, Allen LA, McIlvennan CK, Rich J, Yancy C, Lee CS, Denfeld QE, Kiernan M, Walsh MN, Adler E, Ruo B, Stehlik J, Kirklin JK, Bedjeti K, Cella D, Hahn EA. Novel measures to assess ventricular assist device patient-reported outcomes: Findings from the MCS A-QOL study. J Heart Lung Transplant. 2024 Jan;43(1):36-50. doi: 10.1016/j.healun.2023.08.007. Epub 2023 Aug 15. PMID 37591454
- [Derived] Hahn EA, Walsh MN, Allen LA, Lee CS, Denfeld QE, Teuteberg JJ, Beiser DG, McIlvennan CK, Lindenfeld J, Klein L, Adler ED, Stehlik J, Ruo B, Bedjeti K, Cummings PD, Vela AM, Grady KL. Validity of Patient-Reported Outcomes Measurement Information System Physical, Mental, and Social Health Measures After Left Ventricular Assist Device Implantation and Implications for Patient Care. Circ Cardiovasc Qual Outcomes. 2023 Feb;16(2):e008690. doi: 10.1161/CIRCOUTCOMES.121.008690. Epub 2023 Feb 8. PMID 36752104
- [Derived] Carroll AJ, Hahn EA, Grady KL. Research engagement and experiences of patients pre- and post-implant of a left ventricular assist device from the mechanical circulatory support measures of adjustment and quality of life (MCS A-QOL) study. Qual Life Res. 2022 Aug;31(8):2457-2470. doi: 10.1007/s11136-022-03111-4. Epub 2022 Mar 8. PMID 35258804